CLINICAL TRIAL: NCT00836199
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Assess Efficacy, Immunogenicity and Safety of 3'-Aminomethylnicotine-P. Aeruginosa r-Exoprotein A Conjugate Vaccine (NicVAX) as an Aid to Smoking Cessation
Brief Title: NicVAX/Placebo as an Aid for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nabi-4514; NIH grant # 1 RC2 DA028837-01
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Smoking Cessation; Smoking; Tobacco Cessation
Keywords: smoking cessation; NicVAX; smoking vaccine; smoking abstinence; smoking; tobacco cessation
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo vaccine (Placebo Comparator)
  Interventions: Biological: Placebo vaccine
- NicVAX vaccine (Experimental)
  Interventions: Biological: NicVAX vaccine

INTERVENTIONS:
Biological: NicVAX vaccine — NicVAX vaccine given 6 times over 6 months
  Arms: NicVAX vaccine
Biological: Placebo vaccine — Placebo vaccine given 6 times over 6 months
  Arms: Placebo vaccine

SUMMARY:
The purpose of this study is to evaluate NicVAX as an aid to smoking cessation for long term abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker who smokes at least 10 cigarettes a day during the past year and wants to quit smoking.
* Smokers who are in good general health.

Exclusion Criteria:

* Prior exposure to NicVAX or any other nicotine vaccine.
* Use of systemic steroids.
* Cancer or cancer treatment in last 5 years.
* HIV infection.
* History of drug or alcohol abuse or dependence within 12 months.
* Significant cardiovascular, hepatic, renal, psychiatric and/or respiratory disease.
* Inability to fulfill all visits for approximately 52 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evaluate NicVAX as an aid to smoking cessation for long term abstinence. | one year

SECONDARY OUTCOMES:
Evaluate abstinence rates at multiple intervals | multiple time points
Evaluate safety and immunogenicity | mulitple time points
Evaluate withdrawal symptoms, smoking satisfaction, cigarette consumption and nicotine dependence. | multiple time points

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Nabi Biopharmaceuticals
Locations (22):
- United States (22):
  - NicVAX Investigator, Tucson, Arizona
  - NicVAX Investigator, Los Angeles, California
  - NicVAX Investigator, Newport Beach, California
  - NicVAX Investigator, San Diego, California
  - NicVAX Investigator, Denver, Colorado
  - NicVAX Investigator, Farmington, Connecticut
  - NicVAX Investigator, Miami, Florida
  - NicVAX Investigator, St. Petersburg, Florida
  - NicVAX Investigator, Boise, Idaho
  - NicVAX Investigator, Lexington, Kentucky
  - NicVAX Investigator, Baltimore, Maryland
  - NicVAX Investigator, College Park, Maryland
  - NicVAX Investigator, Boston, Massachusetts
  - NicVAX Investigator, Minneapolis, Minnesota
  - NicVAX Investigator, Omaha, Nebraska
  - NicVAX Investigator, Rochester, New York
  - NicVAX Investigator, Raleigh, North Carolina
  - NicVAX Investigator, Portland, Oregon
  - NicVAX Investigator, Draper, Utah
  - NicVAX Investigator, Norfolk, Virginia
  - NicVAX Investigator, Seattle, Washington
  - NicVAX Investigator, Madison, Wisconsin

REFERENCES:
- [Derived] Fahim RE, Kessler PD, Fuller SA, Kalnik MW. Nicotine vaccines. CNS Neurol Disord Drug Targets. 2011 Dec;10(8):905-15. doi: 10.2174/187152711799219343. PMID 22229310